CLINICAL TRIAL: NCT06876597
Title: Motor-Cognitive Interactive Upper Limb Rehabilitation Robot Intervention for Post-Stroke Motor Dysfunction: A Multicenter Randomized Controlled Study
Brief Title: Motor-Cognitive Interactive Upper Limb Robot Rehabilitation for Post-Stroke Motor Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lidian Chen (Other)
Collaborators: Fujian University of Traditional Chinese Medicine Affiliated Rehabilitation Hospital (Unknown); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); China Rehabilitation Research Center (Other Government); Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong, China (Unknown); Shanghai Sunshine Rehabilitation Center (Unknown)
Responsible Party: Sponsor-Investigator, Lidian Chen, Professor, Fujian University of Traditional Chinese Medicine
Organization: Fujian University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FujianUTCM-3
Record Dates: First submitted 2025-02-19; First posted 2025-03-14 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-02

CONDITIONS: Stroke
Keywords: upeer; motor-cognitive interaction; robot
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor-cognitive interactive robot-assisted training (Experimental)
  Interventions: Device: Motor-cognitive interactive robot
- Motor-focused robot-assisted training (Experimental)
  Interventions: Device: Motor-focused robot
- Conventional rehabilitation training (Experimental)
  Interventions: Behavioral: Conventional rehabilitation training

INTERVENTIONS:
Device: Motor-cognitive interactive robot — Motor-cognitive interactive robot-assisted training integrates motor and cognitive rehabilitation using an upper limb rehabilitation robot. If patients cannot actively lift the robotic arm, an eye-tracking mode detects movement intention and guides the arm along predefined trajectories, adjusting motor and cognitive loads dynamically. As motor function improves, training shifts to an active mode with increased resistance. Patients complete cognitive tasks before moving the robotic arm, while the system monitors movement parameters and provides real-time feedback. Training consists of 60-minute sessions, five days per week for four weeks. Motor load progresses by increasing robotic arm speed or resistance, while cognitive load advances based on task accuracy, ensuring personalized and adaptive rehabilitation.
  Arms: Motor-cognitive interactive robot-assisted training
Device: Motor-focused robot — Motor-focused robot-assisted training primarily emphasizes motor rehabilitation through the use of an upper limb rehabilitation robot. When patients are unable to actively lift the robotic arm, an eye-tracking mode is employed to guide movements, with adjustments made solely to the motor load. As motor function improves, the training transitions to an active mode, progressively increasing resistance while maintaining a constant, minimal level of cognitive difficulty. Patients are required to complete cognitive tasks before initiating movement of the robotic arm, while the system monitors key movement parameters and provides real-time feedback. Training consists of 60-minute sessions, five days per week for four weeks. Motor load is progressively increased by adjusting the speed or resistance of the robotic arm, while cognitive load remains consistently at the lowest level throughout the training.
  Arms: Motor-focused robot-assisted training
Behavioral: Conventional rehabilitation training — Conventional rehabilitation training adheres to internationally established guidelines and employs task-oriented approaches tailored to activities of daily living (ADLs). The therapeutic regimen incorporates fundamental motor skill exercises, including but not limited to grasp-and-release maneuvers, targeted reaching, fine motor skill development (e.g., button manipulation, zipper operation), and bilateral coordination tasks (e.g., garment folding, towel wringing). The intervention protocol emphasizes progressive task difficulty and functional task integration, with each session lasting 60 minutes. The treatment schedule consists of daily sessions, five times per week, over a four-week duration.
  Arms: Conventional rehabilitation training

SUMMARY:
This study aims to investigate the effects of motor-cognitive interactive robot-assisted training on improving upper limb motor dysfunction after stroke. By observing different combinations of motor and cognitive components in the training, the study will clarify the relationship between the proportion of motor and cognitive elements and the recovery of upper limb motor function. The goal is to optimize the training protocol for upper limb rehabilitation robots and enhance their therapeutic outcomes.

Participants will be randomly assigned to one of three groups: motor-cognitive interactive robot-assisted training, motor-focused robot-assisted training, or conventional rehabilitation training. Training sessions will last 60 minutes, occur 5 times per week, and continue for 4 weeks. Researchers will measure changes in upper limb function and monitor for any adverse events during the training.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of stroke confirmed by CT or MRI.
2. Age between 40 and 80 years, with no gender restrictions.
3. First-ever stroke with unilateral limb paralysis.
4. Onset of stroke between 2 weeks and 6 months prior, with an FMA-UE score of 8-44.
5. Willingness to participate and provide written informed consent.

Exclusion Criteria:

1. History of neuromuscular diseases, malignant tumors, or other severe uncontrolled conditions, including cardiac, renal, or hepatic diseases.
2. Seated balance score < 2, or inability to maintain a sitting position for more than 60 minutes.
3. Modified Ashworth Scale score > 2.
4. Visual Analog Scale (VAS) score > 3 for hemiplegic shoulder pain.
5. Boston Diagnostic Aphasia Examination score < 3.
6. Severe visual impairment preventing participation in upper limb robot-assisted rehabilitation training.
7. Hamilton Depression Scale score >17, indicating moderate to severe depressive symptoms.
8. Participation in other clinical trials that may interfere with the results of this study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1047 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity Scale | 4 weeks (post-intervention)
  Score range 0-66, higher scores indicate better upper limb motor recovery.

SECONDARY OUTCOMES:
Fugl-Meyer Upper Extremity Scale | 3 months (post-intervention follow-up)
  Score range 0-66, higher scores indicate better upper limb motor recovery.
Upper limb kinematics during standardized 3D grid tasks | 4 weeks
  The investigators quantify upper limb kinematics using the robot through standardized 3D grid-pointing tasks to measure motion trajectories during task execution.
Upper Limb Muscle Strength Assessment | 4 weeks, 3 months
  Muscle strength is assessed using Manual Muscle Testing (MMT) graded via the Medical Research Council (MRC) Scale (range: 0-5, where 0 = no muscle contraction and 5 = normal strength, higher scores indicate better outcomes).
Modified Barthel Index | 4 weeks, 3 months
  Score range 0-100, higher scores indicate better independence in activities of daily living.
Montreal Cognitive Assessment | 4 weeks, 3 months
  Score range 0-30, higher scores indicate better cognitive function.
Auditory Verbal Learning Test | 4 weeks, 3 months
Trail Making Test Part A | 4 weeks, 3 months
Trail Making Test Part B | 4 weeks, 3 months
Stroke-Specific Quality of Life Scale | 4 weeks, 3 months
  Score range 49-245, higher scores indicate better health-related quality of life in stroke survivors.

OTHER OUTCOMES:
Exercise-associated Blood Biomarkers | 4 weeks
  Quantitative measurement of exercise-associated biomarkers in venous blood using standardized ELISA kits
Multimodal Neuroimaging Analysis | 4 weeks
  Structural (T1-MPRAGE) and resting-state fMRI data acquired via 3T MRI. Structural analysis includes voxel-based morphometry (VBM) for gray matter volume. Functional analysis covers: ALFF, ReHo, FC, and graph-theory network topology (global/local efficiency).

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian University of Traditional Chinese Medicine, Fuzhou, China

IPD SHARING:
Plan to Share IPD: No